CLINICAL TRIAL: NCT06511258
Title: The STRIVE Before Surgery Pilot Trial: a Vanguard Pragmatic Multicenter Randomized Trial of Structured TRaining to Improve Fitness in a Virtual Environment (STRIVE) Before Surgery
Brief Title: The STRIVE Before Surgery Trial
Acronym: STRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OHSN-REB 20230399-01T
Record Dates: First submitted 2024-06-24; First posted 2024-07-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Surgery-Complications; Disability Physical
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patient-reported outcome assessors will be blinded and abstractors collecting routine data are unaware of allocation.
  To support blinding, improve enrollment and reflect usual care, widely available physical activity (World Health Organization Recommendations for Physical Activity for ages 18-64 and >65) and healthy eating recommendations (Canada's Food Guide Snapshot) documents will be provided to control participants (without active or online support).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation (Experimental): The intervention consists of exercise, nutritional support and breathing techniques. The exercise component consists of 1) strength training; 2) cardio and 3) stretching. Participants will be encouraged to complete self-directed and/or group sessions >= 3 times per week. Each intervention participant will be provided a unique login to the virtual prehabilitation platform, which is the STRIVE Trial website. The nutrition component includes: 1) protein supplementation; 2) nutrition advice to support healthy eating. For the breathing component, participants will be encouraged to watch the video on Inspiratory Muscle Training (IMT) which involves diaphragmatic breathing and coughing/huffing. They will also be provided with an instruction booklet to take to hospital with them to support postoperative conduct of IMT during early recovery.
  Interventions: Behavioral: Prehabilitation
- Control (No Intervention): To support blinding, improve enrollment and reflect usual care, widely available physical activity (World Health Organization Recommendations for Physical Activity for ages 18-64 and >65) and healthy eating recommendations (Canada's Food Guide Snapshot) documents will be provided to control participants (without active or online support).

INTERVENTIONS:
Behavioral: Prehabilitation — The intervention includes 3 aspects (exercise, nutrition and breathing). Our intervention is a home-based multimodal prehabilitation program supported through an online platform.
  Arms: Prehabilitation

SUMMARY:
The STRIVE Before Surgery Trial evaluates patient-reported disability at 30 days after surgery following participating in a home-based multimodal prehabilitation program supported through an online platform. Half of the participants will be randomized into the prehabilitation group, while the other half will be randomized into the control group.

DETAILED DESCRIPTION:
Background: The number of people presenting for surgery, and their risk profile, are increasing. People presenting for surgery face substantial risk of postoperative adverse events. Fifteen to 30% of patients suffer a serious medical or surgical complication after surgery, and 1 in 5 develop a new patient-reported disability that reflects a loss of independence in day-to-day life. More than 1.4 million inpatient surgical procedures are performed in Canada each year. Globally, >300 million surgical procedures occur annually. As an increasing number of people present for surgery, the average risk profile of this population is rising. Surgical patients are typically older and live with comorbidity. This means that strategies to improve patient outcomes and reduce resource utilization are urgently needed. Patients, the public, clinicians, and policy makers participating in 2 separate James Lind Alliance Priority Setting Partnerships (Canada & UK) identified prehabilitation as a Top 10 priority for perioperative research. Furthermore, prehabilitation is currently discussed in the popular media as a strategy to improve outcomes for the growing number of high-risk patients presenting for surgery.

Overarching Aim: The pilot phase evaluated three pragmatic elements (recruitment, adherence, and follow-up) that our experience in prehabilitation research demonstrate are necessary to support successful, large-scale evaluation. Data from the pilot phase will be combined with this full-scale trial. The full-scale trial will evaluate patient reported disability at 30 days after surgery.

Methods:

Design, setting and participants: The STRIVE Before Surgery Trial is an assessor blinded multicenter individual patient parallel-arm vanguard pragmatic randomized controlled trial.

People => 18 years old having inpatient abdominal, thoracic, pelvic, head-and-neck or vascular surgery with expected length of stay of => 2 days will be included.

Intervention: The intervention includes 3 aspects (exercise, nutrition and breathing). Our intervention is a home-based multimodal prehabilitation program supported through an online platform.

Outcomes and sample size: Primary outcome is patient-reported disability 30 days after surgery. Secondary outcomes are days at home in the 30 days after surgery, survival, health-related quality of life, length of stay, patient safety indicators, intensive care unit admission, non-home discharge, readmission, emergency department visits, health system costs, and elicitation of patient, clinician and researcher-identified barriers to our pragmatic trial using the Theoretical Domains Framework. Our trial sample size calculation is informed by parameter estimates from the pilot phase. A sample of 902 patients (451 per arm) will provide 90% power to detect a 5% minimally important difference between the mean WHODAS scores using an F-test from an Analysis of Covariance (ANCOVA) at the two-sided 5% significance level. We conservatively assumed a common standard deviation of 23 (equal to the upper limit of the 95% CI observed in our vanguard trial) and a correlation with baseline of 0.3. We also allowed for up to 10% attrition.

Expertise: The team features multidisciplinary clinical and methodological experts, nationally representative knowledge users and patient representatives.

Expected outcomes: Despite systematic review findings that exercise prehabilitation may improve physical performance and function, limitations exist that preclude generalizability, including many identified studies being high or unclear risk of bias and single center studies with <100 participants. The investigators aim to conduct this low risk of bias, mutli-center study of adult surgical patients >18 years to address this gap.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Scheduled, or on the pathway, for inpatient abdominal, thoracic, pelvic, head-and-neck or vascular surgery
3. Expected surgery date between 3 and 12 weeks from enrollment
4. Valid provincial health insurance number
5. Access to internet-enabled device
6. Email address

Exclusion Criteria:

1. Inability to read and communicate in English
2. Cognitive impairment preventing ability to provide informed consent independently
3. No telephone/cell phone
4. Cardiac, neurological or orthopedic procedure
5. Surgery with no curative intent (palliative surgery)
6. Patient not interested in participating in the context of their TAPA score
7. Any of the following cardiovascular conditions:

   1. Severe valvular heart disease that limits a patient's ability to ambulate on level ground, or is associated with syncope or dyspnea
   2. Severe cardiac dysrhythmias that limit a patient's ability to ambulate on level ground, or is associated with syncope or dyspnea
   3. Recent myocardial infarction (within 6 weeks prior to enrollment - based on the Heart and Stroke Foundation's HeartWalk program)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 902 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2031-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported disability using the World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | 1 month
  The WHODAS is a patient-reported disability scale that assesses limitations in six major life domains (i.e., cognition, mobility, self-care, social interaction, life activities, participation in society). Each questionnaire item is scored on a Likert scale ranging from 0 to 4. The sum of the responses is the WHODAS Disability Score (range: 0 to 48), which is expressed as a percentage of the maximum possible score

SECONDARY OUTCOMES:
EuroQol Quality of Life Scale (EQ-5D-5L) | 1 month, 3 months, 1 year
  This is a well-validated instrument with Canadian valuation statistics and national implementation used to measure health-related quality of life after surgery and to inform incremental cost per quality-adjusted life year gained. Participants are asked to select one answer under each domain (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Responses range from having no problems with a particular domain to being unable to engage in that particular domain. Participants are asked to identify on a scale of 0-100 how good or bad their health is on that given day (0 being worst health they can imagine, 100 being best health they can imagine).
A count of days at home in the 30-days after surgery | 1 month
  Count of days at home in the 30-days after surgery is a validated patient-centered outcome that can be ascertained from routinely collected data
Survival | 1 month, 1 year
  All cause deaths and survival time in the 30-days and year after surgery will be captured from vital statistics
Length of stay | 1 year
  Days from surgical admission to discharge will be calculated
Details of patient safety indicators | 1 year
  A validated set of in-hospital patient safety indicators will be captured from the index hospitalization record
Intensive care unit (ICU) admissions | 1 year
  ICU admissions will be accurately captured by administrative data
Intensive care unit (ICU) length of stay | 1 year
  ICU length of stay will be accurately captured by administrative data
Non-home discharge | 1 year
  Discharge from the index hospitalization via transfer to a non-home location or death will be captured
Count of readmissions | 1 month
  Count of any acute hospitalization in the 30-days after surgery
Time to first readmission | 1 month
  Time to first acute hospitalization in the 30-days after surgery
Time to first emergency department visit | 1 month
  Time to first emergency department visit in the 30-days after surgery.
Count of emergency department visits | 1 month
  Count of any emergency department visits in the 30-days after surgery.
Health system costs | 1 month, 1 year
  A validated patient-level costing algorithm will be used to capture all health system costs accrued within 30-days and 1-year after surgery
Elicitation of patient, clinician and researcher-identified barriers to our pragmatic trial using the Theoretical Domains Framework | 1 year
  For each target group, the frequency of domains identified as barriers will be calculated
In-hospital Complications | up to 1 month
  Postoperative Morbidity Survey (POMS) is a tool used to identify complications. At time of discharge, participants will be administered a patient-reported version of the POMS tool.
Patient-reported disability using the World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | 3 months, 1 year
  The WHODAS is a patient-reported disability scale that assesses limitations in six major life domains (i.e., cognition, mobility, self-care, social interaction, life activities, participation in society). Each questionnaire item is scored on a Likert scale ranging from 0 to 4. The sum of the responses is the WHODAS Disability Score (range: 0 to 48), which is expressed as a percentage of the maximum possible score

CONTACTS AND LOCATIONS:
Overall Officials: Daniel McIsaac, MD,MPH,FRCPC, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, including data dictionaries, will be available. This includes individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). The Study Protocol, Statistical Analysis Plan and Informed Consent Form will also be made available. Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data. Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to the Principal Investigator. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.
Supporting Information: SAP
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to the Principal Investigator. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.